CLINICAL TRIAL: NCT01123577
Title: Evaluation of Integrating Self Blood Pressure Monitoring Into Urban Primary Care Practices to Improve Ethnic/ Racial Disparities in Hypertension
Brief Title: Evaluation of Integrating Self Blood Pressure Monitoring Into Urban Primary Care Practices
Acronym: ESBPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Department of Health and Mental Hygiene (Other Government)
Collaborators: Robert Wood Johnson Foundation (Other); NYU Langone Health (Other); Riverdale Family Practice, New York City (Unknown); Heritage Health Center (HHHNYC), New York City (Unknown)
Responsible Party: Principal Investigator, Stella Yi, Principal Investigator, New York City Department of Health and Mental Hygiene
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCIP-CVD-ESBPM2010
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Hypertension; Cardiovascular Disease
Keywords: Self Blood Pressure Monitoring; SBPM; Randomized Control Trial; Hypertension (HTN); Cardiovascular Disease (CVD); HTN; CVD
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Home Blood Pressure Monitor Group
- Control (No Intervention): Participants receive usual care by providers.

INTERVENTIONS:
Other: Home Blood Pressure Monitor Group — Participants receive home monitors, modems, educational materials and training. Participants will send home BP readings to research database monthly and receive usual care by providers for 9 months.
  Arms: Intervention

SUMMARY:
Background:

Hypertension (HTN) is a major risk factor for cardiovascular disease (CVD), the leading cause of death in the United States and New York City (NYC). One in 4 NYC adults has hypertension, with higher prevalence in both Blacks and Latinos compared to Whites (Angell 2008). In NYC, only 65% of all adults with HTN and on treatment are controlled (Angell 2008).

Self-blood pressure monitoring (SBPM) is associated with reduced blood pressure in patients with hypertension (Cappuccio 2004). Studies suggest that SBPM may increase control either by inducing clinicians to titrate medication more actively, (Agency for Healthcare Research and Quality 2002) by engaging patients to participate in their own health care, (Taylor 2007) or a combination of the two.

However, minimal research has been done to evaluate the effectiveness of SBPM in different racial and/or ethnic groups or in low income populations or to discern effective patterns of SBPM use by patients. Best practices for integration of self monitoring into HTN into regular treatment have also yet to be established.

Objectives:

The goal of this study is to assess the impact of SBPM under conditions consistent with existing community health clinic resources and infrastructure in NYC's medically underserved neighborhoods using commonly available automated home BP monitors. By using a community clinic's electronic health record (EHR) and automated BP monitors with the capability to transmit readings to a research database, we can facilitate a more rigorous evaluation of a pilot SBPM intervention and assess patterns of home monitor use and clinical management and their association with outcomes.

The three specific aims of this intervention are to:

1. Assess whether use of SBPM reduces elevated BP and increases HTN control to similar levels in two historically understudied minority populations, Blacks and Latinos.
2. Confirm pilot findings by assessing the impact of SBPM on BP and HTN control compared to usual care using randomized controlled trial methodology.
3. Develop standards and refine guidance for the effective use of SBPM that can be easily communicated to key stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients attending one of the participating primary care clinics
* Diagnosis of hypertension for at least 6 months
* Ethnicity or Race of Latino, Black or White
* Physically and mentally able to monitor BP at home
* *Uncontrolled BP at last office visit
* *Uncontrolled BP at current office visit

Note: *Uncontrolled BP is defined as systolic BP ≥ 140 and/or diastolic BP ≥ 90, or systolic BP ≥ 130 and/or diastolic BP ≥ 80 mm Hg for participants with chronic kidney disease or diabetes.

Exclusion Criteria:

* Arm circumference greater than 17.5 inches (maximum size of large BP cuff)
* Already monitoring BP at home at request of health care provider
* No access to a land line telephone line (to upload home readings)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 899 (Actual)
Dates: Start 2010-05; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Absolute and relative changes in systolic and diastolic BP in the intervention and control groups. | 9 months
Proportion of intervention participants achieving BP control compared to control participants | 9 months
Trajectory of BP changes over time. | 9 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Lutheran Family Health Centers, Brooklyn, New York
  - New York City Department of Health and Mental Hygiene, New York, New York
  - Heritage Health Care, New York, New York
  - Riverdale Family Practice, The Bronx, New York

REFERENCES:
- [Background] Cappuccio FP, Kerry SM, Forbes L, Donald A. Blood pressure control by home monitoring: meta-analysis of randomised trials. BMJ. 2004 Jul 17;329(7458):145. doi: 10.1136/bmj.38121.684410.AE. Epub 2004 Jun 11. PMID 15194600
- [Background] Angell SY, Garg RK, Gwynn RC, Bash L, Thorpe LE, Frieden TR. Prevalence, awareness, treatment, and predictors of control of hypertension in New York City. Circ Cardiovasc Qual Outcomes. 2008 Sep;1(1):46-53. doi: 10.1161/CIRCOUTCOMES.108.791954. PMID 20031787
- [Background] Taylor JR, Campbell KM. Home monitoring of glucose and blood pressure. Am Fam Physician. 2007 Jul 15;76(2):255-60. PMID 17695570
- [Background] Agency for Healthcare Research and Quality. Utility of Blood Pressure Monitoring Outside the Clinic Setting: Agency for Healthcare Research and Quality; 2002.
- [Derived] Yi SS, Tabaei BP, Angell SY, Rapin A, Buck MD, Pagano WG, Maselli FJ, Simmons A, Chamany S. Self-blood pressure monitoring in an urban, ethnically diverse population: a randomized clinical trial utilizing the electronic health record. Circ Cardiovasc Qual Outcomes. 2015 Mar;8(2):138-45. doi: 10.1161/CIRCOUTCOMES.114.000950. Epub 2015 Mar 3. PMID 25737487